CLINICAL TRIAL: NCT06071260
Title: Short-term Effects of 0.01% Atropine on Adult Myopes Pupil Size and Subjective Quality of Vision
Brief Title: Effect of Atropine on Pupil Size and Quality of Vision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Atropine2023-2
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Myopia, Progressive
Keywords: Myopia; Atropine; Eye drops; Quality of vision; Pupil size
MeSH Terms: conditions — Myopia, Degenerative; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Participants will receive 0.01% atropine (0.1 mg/ml)
  Interventions: Drug: 0.01% atropine eye drop

INTERVENTIONS:
Drug: 0.01% atropine eye drop — One drop of 0.01% atropine will be administered to both eyes before bedtime. Baseline parameters were measured before and after atropine application.
  Other Names: Low concentration atropine

SUMMARY:
This aims to investigated the short-term (12, 16, and 20 h) effects of 0.01% atropine (0.1 mg/ml) on pupil size and subjective quality of vision in participants with myopia. Particpants will receive 0.01% atropine one drop to both eyes before bedtime. Baseline parameters were measured before atropine application. Changes in pupil sizes, under photopic and mesopic conditions, high-order aberration, and tear meniscus height were observed over the next day (12, 16, and 20 h).

DETAILED DESCRIPTION:
The utilisation of atropine drops is a common practise in order to induce pupil dilatation, impede accommodation, and decelerate the advancement of myopia. Research findings indicate that the treatment of atropine at a low concentration of 0.01% has been observed to effectively slow down the advancement of myopia, with a reduction rate ranging from 60% to 83%. The administration of a lesser dose of atropine demonstrates a decreased occurrence of undesirable effects in comparison to the administration of atropine at a high concentration of 1.0%. Nevertheless, it is crucial to acknowledge that even when present in low concentrations, atropine still exerts an influence on both pupil size and pupil responsiveness. This investigation employs a prospective cohort study design, in which a set of objective and subjective assessments will be carried out before and after the injection of 0.01% atropine for a duration of 18 hours. The main aim of this study is to determine the effects of a specific concentration of atropine on several factors, including: 1) visual acuity; 2) pupil diameter; 3) subjective perception of vision quality; and 4) intraocular pressure. The objective of this study is to examine the effects of the eye drops on ocular health and determine the degree of patient acceptance about their prospective use as a preventive measure for myopia. The researchers have a positive expectation that the administration of the drops will have minimal influence on the participants in terms of side effects. However, the outcomes of this study will provide valuable insights for children and patients in effectively managing the side effects associated with the use of atropine for myopia control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with myopia
* Able to read and comprehend Chinese and willing to give informed consent as demonstrated by signing a record of informed consent.
* Be between 18 and 60 years old, male or female.
* Willing to apply eye drops once nightly at bedtime for one time and follow the clinical trial visit schedule as directed by the Investigator.
* Willing to answer the questionnaire about subjective measurements.
* Have ocular findings deemed to be myopic.
* No history of wearing contact lens.
* Vision correctable to at least 20/25 or better in each eye with spectacles.

Exclusion Criteria:

* Any pre-existing ocular irritation, injury or condition, including infection or disease.
* Any systemic disease that adversely affects ocular health e.g. diabetes, Graves disease, and auto-immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjögrens syndrome and systemic lupus erythematosus. - - Conditions such as systemic hypertension and arthritis do not automatically exclude prospective participants.
* Use of or a need for concurrent ocular medication at enrolment and/or during the clinical trial.
* Use of or a need for any systemic medication or topical medications which may alter normal ocular findings / are known to affect a participant's ocular health / physiology or contact lens performance either in an adverse or beneficial manner at enrolment and/or during the clinical trial.
* History of eye surgery
* History of use of any myopia control interventions such as Orthokeratology, Rigid Permeable Contact Lenses Eye surgery within 12 weeks immediately prior to enrolment for this trial.
* Currently treated with other interventions for myopia control
* Contraindications to atropine such as pulmonary disease, heart conditions and ADHD
* Known allergy or intolerance to ingredients to atropine eye-drops and other derivatives of anti-muscarinic receptor agents.
* Currently enrolled in another clinical trial.

NB: Systemic antihistamines are allowed on an "as needed basis", provided they are not used prophylactically during the trial and at least 24 hours before the clinical trial product is used.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in pupil size | Baseline (before 0.01% atropine eye drop), 12 hours, 16 hours, and 20 hours.
  Pupil size will be recorded before and after the administration of 0.01% atropine eye drop using the OPD-Scan III (NEIDEK, Japan) device.

SECONDARY OUTCOMES:
Change in subjective quality of vision | Baseline (before 0.01% atropine eye drop), 12 hours, 16 hours, and 20 hours.
  Subjective quality of vision will be recorded before and after the administration of 0.01% atropine eye drop.
Change in high-order aberration | Baseline (before 0.01% atropine eye drop), 12 hours, 16 hours, and 20 hours.
  Change in high-order aberration will be recorded before and after administering 0.01% atropine eye drop using the OPD-Scan III (NEIDEK, Japan) device.

CONTACTS AND LOCATIONS:
Locations (1):
- He Eye Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Background] Sankaridurg PR, Holden BA. Practical applications to modify and control the development of ametropia. Eye (Lond). 2014 Feb;28(2):134-41. doi: 10.1038/eye.2013.255. Epub 2013 Dec 6. PMID 24310242
- [Background] Polling JR, Kok RG, Tideman JW, Meskat B, Klaver CC. Effectiveness study of atropine for progressive myopia in Europeans. Eye (Lond). 2016 Jul;30(7):998-1004. doi: 10.1038/eye.2016.78. Epub 2016 Apr 22. PMID 27101751
- [Background] Chia A, Lu QS, Tan D. Five-Year Clinical Trial on Atropine for the Treatment of Myopia 2: Myopia Control with Atropine 0.01% Eyedrops. Ophthalmology. 2016 Feb;123(2):391-399. doi: 10.1016/j.ophtha.2015.07.004. Epub 2015 Aug 11. PMID 26271839
- [Background] Cooper J, Eisenberg N, Schulman E, Wang FM. Maximum atropine dose without clinical signs or symptoms. Optom Vis Sci. 2013 Dec;90(12):1467-72. doi: 10.1097/OPX.0000000000000037. PMID 24076540